CLINICAL TRIAL: NCT00437840
Title: A Placebo-controlled, Single-blind, Randomised, Human Volunteer Study Investigating the Tolerability and Pharmacokinetics of Escalating Single Oral Doses of GSK598809 in Smokers
Brief Title: A Study To Investigate The Safety, Tolerability And Blood Levels Of GSK598809
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Purpose: Treatment
Other Study IDs: DAN107606
Record Dates: First submitted 2007-02-20; First posted 2007-02-21 (Estimated); Last update posted 2017-08-07 (Actual); Status verified 2017-08

CONDITIONS: Substance Dependence
Keywords: healthy volunteers,; tolerability,; pharmacokinetics,; pharmacodynamics; safety,; smoking,
MeSH Terms: conditions — Substance-Related Disorders; Smoking | interventions — GSK598809

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Treatment Arm A (Experimental): In Arm A dosing subject will receive Placebo in Week 1, 10 milligram (mg) of GSK598809 in Week 2, 25 mg of GSK598809 in Week 3, 75 mg of GSK598809 in Week 4. Subjects will have a wash-out of period of one week before receiving another dose.
  Interventions: Drug: GSK598809; Drug: Placebo
- Treatment Arm B (Experimental): In Arm B dosing subject will receive 10 mg of GSK598809 in Week 1, Placebo in Week 2, 25 mg of GSK598809 in Week 3, 75 mg of GSK598809 in Week 4. Subjects will have a wash-out of period of one week before receiving another dose.
  Interventions: Drug: GSK598809; Drug: Placebo
- Treatment Arm C (Experimental): In Arm C dosing subject will receive 10 mg of GSK598809 in Week 1, 25 mg of GSK598809 in Week 2, Placebo in Week 3, 75 mg of GSK598809 in Week 4. Subjects will have a wash-out of period of one week before receiving another dose.
  Interventions: Drug: GSK598809; Drug: Placebo
- Treatment Arm D (Experimental): In Arm D dosing subject will receive 10 mg of GSK598809 in Week 1, 25 mg of GSK598809 in Week 2, 75 mg of GSK598809 in Week 3, Placebo in Week 4. Subjects will have a wash-out of period of one week before receiving another dose.
  Interventions: Drug: GSK598809; Drug: Placebo

INTERVENTIONS:
Drug: GSK598809 — GSK598809 capsules will be available in dose strength of 5 and 25 mg. Subjects will receive single oral dose of GSK598809 n order to achieve the required dose.
Drug: Placebo — Subjects will receive single oral dose of matching placebo tablet to GSK598809.

SUMMARY:
GSK598809 is being developed to facilitate overcoming an addiction to nicotine and to help people stop smoking. This study will investigate if GSK598809 is safe and tolerated in people who smoke and will also look at blood levels of GSK598809 and nicotine.

ELIGIBILITY:
Inclusion criteria:

* Healthy adult male smoker between the ages of 18 and 50 years
* Body weight greater than 50kg and BMI between 18.5-29.9 kg/m2.
* No abnormalities on the medical, psychiatric or laboratory evaluation
* Smoke on average more than 20 but less that 40 cigarettes per day for the past year and not tried to give up in the 3 months before the study.

Exclusion criteria:

* History of psychiatric disorder or sleep disorder.
* Receiving treatment for smoking cessation.
* Use tobacco products other than cigarettes.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2007-03-20 (Actual); Primary Completion 2007-06-20 (Actual); Study Completion 2007-06-20 (Actual)

PRIMARY OUTCOMES:
Safety measures: ECG, Vital Signs, Adverse Events | for 48 hours after dosing.
PK: Blood levels of GSK598809 and nicotine | for 96 hours after dosing

SECONDARY OUTCOMES:
Questionnaires on nicotine craving | for 24 hours after dosing
Tests on cognition (thinking) | for 48 hours after dosing

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Berlin, Germany

REFERENCES:
- See also: Results for study DAN107606 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/DAN107606?search=study&search_terms=DAN107606#rs